CLINICAL TRIAL: NCT05321524
Title: A Multicenter, Open-Label, Single- and Multiple-Dose, Dose-Finding Study, With an Optional Open-Label Extension to Assess the Safety, Tolerability, and Pharmacokinetics of Obeticholic Acid in Pediatric Subjects With Biliary Atresia
Brief Title: Obeticholic Acid in Pediatric Subjects With Biliary Atresia
Acronym: CARE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After extensive efforts to improve recruitment, it is deemed not feasible to enroll the requisite number of subjects to generate data needed to meet the study objectives. EMA Paediatric Committee agreed with the Sponsor to terminate this study.
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 747-206
Record Dates: First submitted 2022-03-18; First posted 2022-04-11 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; hepatoportoenterostomy (HPE); Kasai portoenterostomy; Liver; Obeticholic Acid
MeSH Terms: conditions — Biliary Atresia | interventions — obeticholic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SD (1.5mg adult-equivalent dose of OCA) + MD Low dose (1.5mg adult-equivalent dose of OCA) (Experimental): At Single Dose (SD) phase, eligible subjects will receive a 1.5 mg adult-equivalent, body weight-based single dose of OCA on Day 1. Enrollment in the Multiple Dose (MD) Phase will occur in a sequential fashion. At Day 28, the first 8 (±1) eligible subjects will be assigned to the Low Dose Cohort and will receive a 1.5 mg adult-equivalent dose of OCA daily for 4 weeks.
  The adult-equivalent dose is based on a 70-kg adult. 2 OCA tablet dose strength (0.1mg and 1.5mg) are available in the study and dose will be determined using weight based dosing chart.
  Interventions: Drug: OCA 0.1mg; Drug: OCA 1.5mg
- SD (1.5mg adult-equivalent dose of OCA) + MD Medium dose (5mg adult-equivalent dose of OCA) (Experimental): At Single Dose (SD) phase, eligible subjects will receive a 1.5 mg adult-equivalent, body weight-based single dose of OCA on Day 1. Upon safety and tolerability assessment in the Low Dose Cohort, 8 (±1) eligible subjects will be assigned to the Medium Dose Cohort and will receive a 5 mg adult-equivalent dose of OCA daily for 4 weeks.
  The adult-equivalent dose is based on a 70-kg adult. 3 OCA tablet dose strength (0.1mg, 1.5mg and 5mg tablets) are available in the study and dose will be determined using weight based dosing chart.
  Interventions: Drug: OCA 0.1mg; Drug: OCA 1.5mg; Drug: OCA 5mg
- SD (1.5mg adult-equivalent dose of OCA) + MD High dose (10mg adult-equivalent dose of OCA) (Experimental): At Single Dose (SD) phase, eligible subjects will receive a 1.5 mg adult-equivalent, body weight-based single dose of OCA on Day 1. Upon safety and tolerability assessment in the Medium Dose Cohort, 8 (±1) eligible subjects will be assigned to the High Dose Cohort and will receive a 10 mg adult-equivalent dose of OCA daily for 4 weeks.
  The adult-equivalent dose is based on a 70-kg adult. 3 OCA tablet dose strength (0.1mg, 1.5mg and 5mg tablets) are available in the study and dose will be determined using weight based dosing chart.
  Interventions: Drug: OCA 0.1mg; Drug: OCA 1.5mg; Drug: OCA 5mg

INTERVENTIONS:
Drug: OCA 0.1mg — Tablets administered orally once daily.
  Other Names: Obeticholic Acid; 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
Drug: OCA 1.5mg — Tablets administered orally once daily.
  Other Names: 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
Drug: OCA 5mg — Tablets administered orally once daily.
  Other Names: 6alpha-ethylchenodeoxycholic acid (6-ECDCA); INT-747
  Arms: SD (1.5mg adult-equivalent dose of OCA) + MD High dose (10mg adult-equivalent dose of OCA); SD (1.5mg adult-equivalent dose of OCA) + MD Medium dose (5mg adult-equivalent dose of OCA)

SUMMARY:
This is a Phase 2, multicenter, open-label, single dose and multi-dose, dose-finding study with an optional open-label extension (OLE) to assess the safety, tolerability, and pharmacokinetics of obeticholic acid (OCA) in pediatric subjects with biliary atresia with successful hepatoportoenterostomy (HPE, also known as a Kasai portoenterosomy). The OLE will continue to evaluate safety, tolerability, pharmacodynamics, and efficacy of OCA. In addition, a change in vitamin A and D levels, and where possible the degree of change in liver stiffness, will be assessed during the OLE.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female pediatric subjects ≥2 to <18 years old
2. Diagnosis of biliary atresia
3. Demonstrated successful HPE (also known as Kasai portoenterostomy) as defined by total bilirubin <2 mg/dL (34.2 μmol/L) at least 3 months post-HPE procedure.
4. Able to swallow tablets (ie, tablet or mini-tablet formulation)

Key Exclusion Criteria:

1. Prior liver transplant or active status on transplant list
2. Conjugated (direct) bilirubin ≥ULN of site specific reference range
3. If conjugated bilirubin is not available: total bilirubin ≥2 mg/dL (34.2 μmol/L)
4. Platelets <150,000/μL
5. INR ≥1.5
6. Current or history of complications of decompensated chronic liver disease including:

   1. high-risk gastroesophageal varices and/or variceal bleeding
   2. clinically evident ascites related to portal hypertension
   3. hepatic encephalopathy
   4. prior placement of portosystemic shunt
   5. hepatopulmonary syndrome or portopulmonary hypertension
   6. hepatorenal syndrome
7. Current intractable pruritus or requires systemic treatment for pruritus within 3 months of Screening (e.g., with bile acid sequestrants or rifampicin)
8. Height and weight Z-score <-2 per site specific ranges
9. Acholic (pale) stools
10. AST >4x ULN
11. ALT >4x ULN
12. GGT >500 U/L
13. Anticoagulation therapy
14. Albumin <3.5 g/dL
15. Ongoing current cholangitis
16. Choledochal cystic disease
17. Renal disease defined as serum creatinine >ULN for subject's age, prior to enrollment

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by the incidence of treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs) | Day 1, 21, and 56.
The plasma concentration of OCA and its conjugates (glyco-OCA and tauro-OCA) | Day 1, 21, and 56.
  Change in plasma concentrations of unconjugated OCA and its conjugates (glyco-OCA and tauro-OCA) will be quantitated, and total OCA concentration will be calculated in the SD and MD Phase.

SECONDARY OUTCOMES:
Biomarkers of FXR-activation: change from baseline of the plasma value of Fibroblast Growth Factor-19 (FGF-19) | Day 1, 21, and 56
Biomarkers of FXR-activation: change from baseline of the plasma value of 7-hydroxyl-4-cholesten-3-one (C4) | Day 1, 21, and 56
Biomarkers of FXR-activation: change from baseline of the plasma value of Endogenous Bile Acids | Day 1, 21, and 56
Biomarkers of hepatobiliary function: Alkaline Phosphatase (ALP) | Time Frame: Day 1, 21, and 56
Biomarkers of hepatobiliary function: Aspartate Aminotransferase (AST) | Time Frame: Day 1, 21, and 56
Biomarkers of hepatobiliary function: Alanine Aminotransferase (ALT) | Time Frame: Day 1, 21, and 56
Biomarkers of hepatobiliary function: Gamma-Glutamyl Transpeptidase (GGT) | Time Frame: Day 1, 21, and 56

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Szczech, MD, Study Director — Intercept Pharmaceuticals
Locations (17):
- Clinques University Saint-Luc, Brussels, Belgium
- France (4):
  - CHU Lille, Lille, ME
  - Hopital de la Timone, Marseille, PACA
  - APHP- Hopital Necker Enfants Malades, Paris
  - CHU de Toulouse Purpan-Hopital des Enfants, Toulouse
- Hannover Medical School, Children's Hospital, Paediatric Gastroenterology and Hepatology,, Hanover, Lower Saxony, Germany
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Shaare-Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
- Italy (2):
  - Centre for Paediatric Hepatology, Bergamo
  - Regina Margherita Children's Hospital, Turin
- University Medical Center Gröningen-Beatrix, children's Hospital, Groningen, Netherlands
- Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Poland
- Spain (2):
  - Passeig Vall d'Hebron, Barcelona
  - Hospital Materno-Infantil de Malaga, Málaga
- Birmingham Children's Hospital, Birmingham, West Midlands, United Kingdom